CLINICAL TRIAL: NCT05720455
Title: A Phase IV, Open Label, Clinical Trial to Assess Safety and Efficacy of Fexofenadine HCL + Pseudoephedrine HCL Fixed Dose Combination in Indian Participants With Allergic Rhinitis (AR) Who Are 12 Years and Above (FAST Trial)
Brief Title: Study to Assess Safety and Efficacy of Fexofenadine Hydrochloride (HCL) + Pseudoephedrine HCL Fixed Dose Combination in Indian Male and Female Participants With Allergic Rhinitis (AR) Who Are 12 Years and Above
Acronym: FAST
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS17348; U1111-1277-6766 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Rhinitis Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — fexofenadine; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fexofenadine HCL + pseudoephedrine HCL (Experimental): Participants will take a tablet containing fexofenadine 60 mg and pseudoephedrine 120 mg twice daily for 10 days (+/- 3 days based on investigator's clinical judgement)
  Interventions: Drug: Fexofenadine HCL and pseudoephedrine HCL

INTERVENTIONS:
Drug: Fexofenadine HCL and pseudoephedrine HCL — Extended-Release Tablets
  Other Names: ALLEGRA® D

SUMMARY:
This is a single group, Phase IV clinical trial to assess the safety and effectiveness of Allegra® D. This study will be conducted in participants with allergic rhinitis who are 12 years of age and above. The individual study duration for each participant would be approximately 16 days (maximum of 13 days intervention + a 3-day post intervention observation). There would be 4 study visits in which the last visit can be done either telephonically or on site. Safety events would be captured for the entire study duration. In addition, the effectiveness of the study drug would be assessed using Nasal symptom score (NSS) and Total symptom score (TSS).

DETAILED DESCRIPTION:
The individual study duration for each participant would be approximately 16 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant (male or female) must be 12 years or more, at the time of signing the informed consent.
* Female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:

  i) Not a woman of childbearing potential (WOCBP) OR ii) A WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 3 days after the last dose of study intervention
* Male participants who agree to follow the contraceptive guidance during the intervention period and for at least 3 days after the last dose of study intervention
* Capable of giving signed informed consent:

  i) Signed informed consent (for participants who are 18 years old or above) ii) Participant assent and parental/legal guardian consent (for participants who are less than 18 years old)

Exclusion Criteria:

* Participants with nasal diseases (hypertrophic rhinitis, paranasal sinusitis, nasal polyps, acute rhinitis, deviation of the nasal septum, etc.), upper respiratory tract infection or acute otitis media that could interfere with judgment of the efficacy of the investigational product (IP) and participants developing cold-like symptoms 30 days before the screening visit
* Participants with severe asthma, bronchiectasis
* Participants using following drugs:

  a) within 5 days prior to the day of screening: i) Intranasal or oral: antiallergic drugs, decongestants, antihistamines, anticholinergic agents, vasoconstrictor, antihistamine-containing cold remedies, agents that can be expected to have an antiallergic/antihistaminic effect, and other agents that are indicated for allergic symptoms (sneezing, rhinorrhea, nasal congestion, etc.) ii) agents that may affect the blood concentration of fexofenadine (macrolide antibiotics, azole fungicides, and preparations containing aluminum hydroxide / magnesium hydroxide) b) within 2 weeks prior to screening visit: i) participants using steroids, sodium cromoglycate/nedocromil or leukotriene modifiers ii) participants receiving monoamine oxidase (MAO) inhibitor therapy iii) participants receiving immunotherapy or immunosuppressants or nonspecific alternative therapy (histamine containing gamma globulin preparations etc)
* Participants who are participating in another study or who have previously participated in another study within the previous 3 months prior to the day of screening
* Participants were excluded from the study if they had hypersensitivity to, fexofenadine HCL, or pseudoephedrine HCL

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2025-06-06 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Day 1 to Day 16
  A TEAE is defined as any adverse event (AE) that occur in between the first investigational medicinal product (IMP) administration (on Day 1) and Day 16.
Number of participants with treatment-emergent serious adverse events (SAEs) | Day 1 to Day 16
  A treatment-emergent SAE is defined as any SAE that occur in between the first investigational medicinal product (IMP) administration (on Day 1) and Day 16.

SECONDARY OUTCOMES:
Mean change from baseline in Total Symptom Score (TSS) | Day 1, Day 13
  The TSS is the sum of physician-assessed nasal symptom scores for sneezing; rhinorrhea; itchy nose, palate, and/or throat; itchy, watery eyes; and nasal congestion, each accessed on 0-4 categorical scale (where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms and 4 = very severe symptoms). Higher score indicated more severe symptoms.
Mean change from baseline in Nasal Congestion Score (NCS) | Day 1, Day 13
  Nasal congestion was assessed by the physician on a 0-4 categorical scale, where 0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms and 4 = very severe symptoms. Higher score indicated more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org